CLINICAL TRIAL: NCT00500825
Title: Influence of Therapeutic Hypothermia on Resting Energy Expenditure in Patients After Cardiopulmonary Resuscitation
Brief Title: Influence of Therapeutic Hypothermia on Resting Energy Expenditure
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Ulrike Holzinger, Medical University of Vienna
Other Study IDs: 486/2003
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Cardiopulmonary resuscitation; Therapeutic hypothermia; resting energy expenditure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients successfully resuscitated after cardiac arrest undergoing therapeutic hypothermia
  Interventions: Procedure: Measurement of Resting Energy Expenditure

INTERVENTIONS:
Procedure: Measurement of Resting Energy Expenditure — Non-invasive measurement of Resting Energy Expenditure
  Other Names: Deltatrac (Ohmeda)

SUMMARY:
The purpose of this study is the evaluation of the influence of therapeutic hypothermia on resting energy expenditure (REE) in patients after cardiopulmonary resuscitation (CPR). We hypothesized that hypothermia would reduce resting energy expenditure in these patients.

DETAILED DESCRIPTION:
Therapeutic hypothermia improves neurologic outcome in patients after cardiopulmonary resuscitation (CPR) because of cardiac arrest. In the present study patients will be cooled to 33 degree Celsius after CPR for 24h. To avoid shivering patients will be analgosedated and medically paralysed. Analgosedation and relaxation have already shown to reduce oxygen consumption up to 20 % in critically ill patients.

In patients with brain injury, who were cooled to 33 degree Celsius using a cooling meadow REE could be significantly reduced. In critically ill patients with pyrexia cooling using a cooling meadow REE could be reduced. Oxygen consumption was reduced about 14,7% per degree Celsius.

So far no studies evaluating influence of therapeutic hypothermia on REE in patients after CPR have been published. Therefore we plan to measure REE in 25 cooled patients after CPR using indirect Calorimetry (Deltatrac II Metabolic Monitor, Datex Instrumentarium, Helsinki, Finland).

ELIGIBILITY:
Inclusion Criteria:

* St.p. CPR
* Indication for therapeutic hypothermia for 24h (33 degrees Celsius)

Exclusion Criteria:

* Contraindication for therapeutic hypothermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Vienna
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2005-07; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Holzinger, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Holzinger U, Brunner R, Losert H, Fuhrmann V, Herkner H, Madl C, Sterz F, Schneeweiss B. Resting energy expenditure and substrate oxidation rates correlate to temperature and outcome after cardiac arrest - a prospective observational cohort study. Crit Care. 2015 Mar 29;19(1):128. doi: 10.1186/s13054-015-0856-2. PMID 25888299